CLINICAL TRIAL: NCT04158323
Title: Survey on the Current Significance of the Flexible Endoscopy as the Gold Standard for Airway Management in Patients With Anticipated Difficult Airway
Brief Title: What is the Gold Standard of Airway Management in the Anticipated Difficult Airway
Acronym: FOI
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: JohannesGUF
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Airway Morbidity
Keywords: flexible endoscopy; awake intubation
MeSH Terms: interventions — Airway Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Airway Management in patients with a anticipated difficult airway — survey of anesthesists and intensive care physician of the perfomans with the flexible endoscope in patients with a anticipated difficult airway

SUMMARY:
A prospective Observationalstudie to analyze the current significance of the awake flexible endoscopy in German hospitals.

DETAILED DESCRIPTION:
The aim of the study is to analyze the current significance of the awake flexible endoscopy in German hospitals, to identify strategies to securing the airway in patients with a anticipated difficult airway. The participants complete a pre-prepared questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* experience in anesthesia or intensive care

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: anesthesists and intensive care physicians
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-11-23 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
What is the current practice for Airway Management in patients with a anticipated difficult airway? | through study completion, an average of 10 minutes
  Evaluation of the current practice to secure the airway in patients with a anticipated difficult airway

SECONDARY OUTCOMES:
What is the most preferred technique for awake flexible endoscopy? | through study completion, an average of 10 minutes
  Evaluation of application (nasal/oral), local anesthestics

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University Medical Center Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany